CLINICAL TRIAL: NCT02499120
Title: A RANDOMIZED, MULTICENTER, DOUBLE-BLIND PHASE 2 STUDY OF PALBOCICLIB PLUS CETUXIMAB VERSUS CETUXIMAB FOR THE TREATMENT OF HUMAN PAPILLOMAVIRUS-NEGATIVE, CETUXIMAB-NAÏVE PATIENTS WITH RECURRENT/METASTATIC SQUAMOUS CELL CARCINOMA OF THE HEAD AND NECK AFTER FAILURE OF ONE PRIOR PLATINUM-CONTAINING CHEMOTHERAPY REGIMEN
Brief Title: Safety And Efficacy Study Of Palbociclib Plus Cetuximab Versus Cetuximab To Treat Head And Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5481044; 2015-000515-41 (EudraCT Number); PALATINUS (Other: Alias Study Number)
Record Dates: First submitted 2015-07-13; First posted 2015-07-15 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Keywords: palbociclib, cetuximab, human papillomavirus, squamous cell carcinoma, head and neck cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell; Head and Neck Neoplasms | interventions — palbociclib; Cetuximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Palbociclib plus Cetuximab (Experimental): Palbociclib, 125 mg, orally once daily (QD) with food on Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle; in combination with Cetuximab, 400 mg/m2 initial dose as a 120-minute IV infusion followed by 250 mg/m2 weekly infused over 60 minutes.
  Interventions: Drug: palbociclib; Drug: Cetuximab
- Placebo plus Cetuximab (Active Comparator): Placebo orally QD with food on Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle; in combination with Cetuximab, 400 mg/m2 initial dose as a 120-minute IV infusion followed by 250 mg/m2 weekly infused over 60 minutes.
  Interventions: Drug: Cetuximab; Drug: Placebo

INTERVENTIONS:
Drug: palbociclib — Palbociclib will be supplied as capsules containing 75 mg, 100 mg, or 125 mg equivalents of palbociclib free base. Administered with food on Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle.
  Other Names: IBRANCE, PD-0332991
  Arms: Palbociclib plus Cetuximab
Drug: Cetuximab — Cetuximab injection for IV infusion will be provided in 100 mg/50 mL, single-use vials, and 200 mg/100 mL, single-use vials. In Japan, cetuximab will be provided in 100 mg/20 mL, single-use vials. Administered, 400 mg/m2 initial dose as a 120-minute IV infusion followed by 250 mg/m2 weekly infused over 60 minutes.
  Other Names: ERBITUX
Drug: Placebo — Placebo for palbociclib will be indistinguishable from the palbociclib capsules and will be supplied as capsules matching in size and color the various palbociclib formulations.
  Administered with food on Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle.
  Arms: Placebo plus Cetuximab

SUMMARY:
The purpose of this study is to determine whether the combination of palbociclib with cetuximab is superior to cetuximab in prolonging overall survival in HPV-negative, cetuximab-naive patients with recurrent/metastatic squamous cell carcinoma of the head and neck.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx, not amenable for salvage surgery or radiotherapy.
* Measurable disease as defined per RECIST v. 1.1. Tumor lesions previously irradiated or subjected to other locoregional therapy will only be deemed measureable if disease progression at the treated site after completion of therapy is clearly documented.
* HPV- negative SCCHN tumor as determined per institutional standard (eg, p16 IHC; multiplex nucleic acid sequence based amplification [NASBA] or other polymerase chain reaction [PCR]-based assays).
* Documented progressive disease according to RECIST v1.1 (Appendix 2) following receipt of at least 2 cycles of one platinum-containing chemotherapy regimen administered for R/M disease (min. 50 mg/m2 for cisplatin, minimum area under the curve [AUC] > 4 for carboplatin).
* Availability of a tumor tissue specimen (ie, archived formalin fixed paraffin embedded tissue [block preferred, or 15 unstained slides]), which will be used for centralized, retrospective biomarker analysis. If archived tumor tissue is not available, then a de novo biopsy will be required for patient participation.

Key Exclusion Criteria:

* Prior nasopharyngeal cancer, salivary gland or sinus tumors.
* More than one chemotherapeutic regimen given for R/M disease. Prior treatment with immunotherapy is allowed.
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases, carcinomatous meningitis, or leptomeningeal disease as indicated by clinical symptoms, cerebral edema, and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated with local therapy (eg, radiotherapy, stereotactic surgery) and are clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization.
* Progressive disease within 3 months after completion of curatively intended treatment for locoregionally advanced SCCHN.
* Difficulty swallowing capsules.
* Prior use of cetuximab in the R/M disease treatment setting (except cetuximab during curative radiotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2018-07-19 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (71):
- United States (14):
  - UC San Diego Medical Center - La Jolla (Thornton Hospital), La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center- Hillcrest, San Diego, California
  - University Medical Center, lnc.:DBA University of Louisville Hospital, Louisville, Kentucky
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - University of Cincinnati Investigational Pharmacy, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UC Health Physicians Office South, West Chester, Ohio
  - Henry Joyce Cancer Clinic, Nashville, Tennessee
- Czechia (5):
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Olomouc, Lekarna, Olomouc
  - Nemocnice Na Bulovce, Centralni laboratore Pavilon c. 8, Prague
  - Nemocnice Na Bulovce, Lekarna, Oddeleni Centralni pripravy, Prague
  - Nemocnice Na Bulovce, Ustav radiacni onkologie, Prague
- Hungary (5):
  - Debreceni Egyetem klinikai Koezpont Onkologiai Intezet, Debrecen
  - Neuro CT Kft, Pécs
  - Pecsi Tudomanyegyetem, Klinikai Kozpont, Laboratoriumi, Pécs
  - Pecsi Tudomanyegyetem, Klinikai Kozpont,, Pécs
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet,Onkologiai Kozpont, Szolnok
- Istituto Nazionale Tumori Napoli, Napoli, Italy
- Japan (4):
  - Aichi cancer center Central hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital/Otolaryngology, Sapporo, Hokkaido
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
- Mexico (6):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Cirugia y Ginecobstetricia de Oaxaca S.A de C.V Hospital Reforma, Oaxaca City, Oaxaca DE Juarez
  - Diaz San Juan Noe, Imagenologia Siglo XXI San Felipe, Oaxaca City, Oaxaca DE Juarez
  - Daniel Javier Mendez Lopez Imagen y Diagnostico Medico IDM, Oaxaca City, Oaxaca DE Juarez
  - Oaxaca Site Management Organization S C, Oaxaca City
- Poland (4):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im. ks. B. Markiewicza, Brzozów
  - Uniwersyteckie Centrum Kliniczne Klinika Onkologii i Radioterapii, Gdansk
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika w Lodzi Oddzial Chemioterapii, Lodz
  - SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie Oddzial Kliniczny Onkologii, Olsztyn
- Romania (5):
  - SC Medisprof SRL, Cluj-Napoca, Cluj
  - Centrul de Oncologie Sf. Nectarie SRL, Craiova, Dolj
  - SC Oncolab SRL, Craiova, Dolj
  - S.C. ONCOCENTER Oncologie Clinica S.R.L., Timișoara, Timiș County
  - Spitalul Clinic Judetean de Urgenta Sibiu, Clinica Oncologie Medicala, Sibiu
- Russia (4):
  - State Budgetary Healthcare Institution of Arkhangelsk Region, Arkhangelsk, Arkhangelskaya oblast
  - State Budgetary Healthcare Institution "Oncology Center #2" of the Ministry of, Sochi, Krasnodarskiy Kray
  - State Autonomous Healthcare Institution Republican Clinical Oncology Dispensary of the Ministry, Kazan', Tatarstan Republic
  - FSBI "National Medical Scientific Centre of Oncology n.a.N.N.Petrov" of the MOH of Russia, Saint Petersburg
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Military Medical Academy, Belgrade
- Slovakia (2):
  - Narodny onkologicky ustav, Bratislava
  - POKO Poprad, s.r.o., Poprad
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (3):
  - Servicio de Oncologia, Pamplona, Navarre
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Cheng Kung University Hospital Department of Pathology, Tainan
  - Tri-Service General Hospital, Taipei
- Ukraine (8):
  - Communal Institution of Kherson Regional Council Kherson Regional Oncological Dispensary, Antonivka, Kherson Oblast
  - Communal Institution "Chernivtsi Regional clinical oncology dispensary",, Chernivtsy
  - SI Dnipropetrovsk Medical Academy of MoH of Ukraine, Chair of Oncology and Medical Radiology, Dnipropetrovsk
  - CI Dnipropetrovsk City Multifunctional Clinical Hospital #4 of Dnipropetrovsk Regional Council, Dnipropetrovsk
  - Regional Clinical Hospital, Department of microsurgery of otolaryngology organs, Ivano-Frankivsk
  - Communal Institution "Krivorizhskiy Oncology Dispensary" of Dnipropetrovsk Regional Council,, Kryvyi Rih
  - Clinic of SI "Institute of Otolaryngology n.a. Prof. O.S. Kolomyichenka of NAMSU", Kyiv
  - Podilskiy Regional Center of Oncology, Chemotherapy Department, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Adkins DR, Lin JC, Sacco A, Ley J, Oppelt P, Vanchenko V, Komashko N, Yen CJ, Wise-Draper T, Lopez-Picazo Gonzalez J, Radulovic S, Shen Q, Thurm H, Martini JF, Hoffman J, Huang X, Melichar B, Tahara M. Palbociclib and cetuximab compared with placebo and cetuximab in platinum-resistant, cetuximab-naive, human papillomavirus-unrelated recurrent or metastatic head and neck squamous cell carcinoma: A double-blind, randomized, phase 2 trial. Oral Oncol. 2021 Apr;115:105192. doi: 10.1016/j.oraloncology.2021.105192. Epub 2021 Feb 8. PMID 33571736
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 125 participants were randomized; among them, 124 participants received study treatments. One (1) participant in the palbociclib + cetuximab treatment group was randomized but not treated.
Groups:
- Palbociclib + Cetuximab: Participants received Palbociclib, 125 mg, orally once daily (QD) with food on Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle in combination with Cetuximab, 400 mg/m^2 initial dose as a 120-minute intravenous (IV) infusion followed by 250 mg/m^2 weekly infused over 60 minutes.
- Placebo + Cetuximab: Participants received Placebo orally QD with food on Day 1 to Day 21 followed by 7 days off treatment in a 28-day cycle in combination with Cetuximab, 400 mg/m^2 initial dose as a 120-minute IV infusion followed by 250 mg/m^2 weekly infused over 60 minutes.
Period: Overall Study
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Started | 65 | 60
Received Treatment | 64 | 60
Completed | 0 | 0
Not Completed | 65 | 60
Not completed — Death | 52 | 43
Not completed — Lost to Follow-up | 1 | 2
Not completed — Participant refused further follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Other | 9 | 10

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab | Total
Number analyzed (Participants) | 65 | 60 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.2) | 60.9 (10.1) | 59.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 57 | 56 | 113
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 46 | 93
  Black | 1 | 1 | 2
  Asian | 15 | 13 | 28
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. OS (in months) was calculated as (date of death - randomization date +1)/30.4. For participants lacking survival data beyond the date of their last follow-up, the OS time was censored on the last date they were known to be alive. Participants lacking survival data beyond randomization had their OS times be censored at randomization. Estimates of OS and its 95% confidence interval were determined using Kaplan-Meier method.
Time Frame: Baseline up to primary completion date (PCD) (about 34 months)
Population: The analysis population was intent-to-treat (ITT) population, which included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 65 | 60
months | 9.7 [7.3 to 13.9] | 7.8 [6.7 to 10.6]
Statistical Analysis 1: Comparison: Palbociclib + Cetuximab vs Placebo + Cetuximab; Test type: Superiority; p = 0.1800, Log Rank — 1-sided p-value was from the log-rank test stratified by stratification factors ECOG(Eastern Cooperative Oncology Group) per randomization; Hazard Ratio (HR) = 0.820, 95% CI 2-sided [0.536 to 1.253]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the date of randomization to the date of the first documentation of objective progression of disease (PD) or death due to any cause, whichever was earlier. Estimates of the PFS curves from the Kaplan Meier method were presented.
Time Frame: Baseline up to PCD (about 34 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 65 | 60
months | 3.9 [3.6 to 5.6] | 4.6 [2.3 to 5.5]
Statistical Analysis 1: Comparison: Palbociclib + Cetuximab vs Placebo + Cetuximab; Test type: Superiority; p = 0.4953, Log Rank — 1-sided p-value was from the log-rank test stratified by stratification factors ECOG per randomization; Hazard Ratio (HR) = 1.000, 95% CI 2-sided [0.669 to 1.495]

3. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR was defined as the overall complete response (CR) or partial response (PR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Objective response rate was defined as the proportion of participants with best overall response (BOR) of CR or PR relative to all randomized.
Time Frame: Baseline up to PCD (about 34 months)
Population: The analysis population was ITT population, which included all participants who were randomized, with study drug assignment designated according to initial randomization, regardless of whether participants received study drug or received a different drug from that to which they were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 65 | 60
Percentage of participants | 27.7 [17.3 to 40.2] | 25.0 [14.7 to 37.9]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit Response (CBR)
Description: CBR was defined as the overall CR, PR, or stable disease>=24 weeks according to the RECIST version 1.1. Clinical benefit response rate was defined as the proportion of participants with CR, PR, or stable disease>= 24 weeks relative to all randomized participants and randomized participants with measurable disease at baseline.
Time Frame: Baseline up to PCD (about 34 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 65 | 60
Percentage of participants | 36.9 [25.3 to 49.8] | 36.7 [24.6 to 50.1]

5. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of disease progression or to death due to any cause, whichever occurred first. If tumor progression data included more than 1 date, the first date was used. DR was calculated as [the date response ended (ie, date of PD or death) - first CR or PR date + 1]/30.4.
Time Frame: Baseline up to PCD (about 34 months)
Population: DR was only calculated for the subgroup of all ITT participants with an objective tumor response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 18 | 15
months | 7.6 [3.7 to 7.7] | 7.4 [3.6 to NA] — Number of participants with confirmed objective response was too small to provide such summary statistics (upper limit of 95% CI).

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events(TEAEs)
Description: AE was defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of the causal relationship to study treatment. TEAEs were defined as AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Causality to study treatment was determined by the investigator. Severity was graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: From the first dose through and including 28 calendar days after the last administration of the study treatment (up to 6.9 years)
Population: The analysis population included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 64 | 60
Participants
  AEs (all causality) | 61 | 56
  AEs (treatment-related) | 58 | 48
  SAEs (all causality) | 25 | 19
  SAEs (treatment-related) | 7 | 2
  Grade 3 or 4 AEs (all causality) | 33 | 19
  Grade 5 AEs (all causality) | 15 | 11
  Grade 3 or 4 AEs (treatment-related) | 34 | 10
  Grade 5 AEs (treatment-related) | 1 | 0

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: The hematology, chemistry and coagulation tests were included in the laboratory examination. Hematology evaluation included hemoglobin, platelets, white blood cell, absolute neutrophils, absolute lymphocytes. Chemistry evaluation included alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen (BUN) or urea, creatinine, uric acid, glucose (non-fasted), albumin, phosphorus or phosphate and hemoglobin A1c (HbA1c). Coagulation evaluation included activated partial thromboplastin time/partial thromboplastin time, international normalized ratio (INR) or prothrombin time.
Time Frame: From the Screening (Day -28) through and including 28 calendar days after the last administration of the study treatment (up to 7 years)
Population: The analysis population included all participants with at least 1 observation of the laboratory test while on study treatment or during lag time.
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 62 | 59
Participants | 61 | 55

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 is a 30 item questionnaire composed of 5 multi-item functional subscales (physical, role, cognitive, emotional, and social functioning), 3 multi-item symptom scales (fatigue, nausea/vomiting, and pain), a global health/quality of life (QOL) subscale, and 6 single items assessing other cancer related symptoms (dyspnea, sleep disturbance, appetite, diarrhea, constipation, and the financial impact of cancer). The questionnaire employed twenty-eight 4 point Likert scales with responses from "not at all" to "very much" and two 7 point Likert scales for global health and overall QOL. For functional and global QOL scales, higher scores represented a better level of functioning and all scores were converted to a 0 to 100 scale. For symptom oriented scales, a higher score represented more severe symptoms, and all scores were converted to a 0-100 scale. Negative changes from baseline indicate deterioration in functioning / global QoL scales and improvement in symptom scales.
Time Frame: Baseline up to PCD (about 34 months)
Population: The analysis population included all ITT participants, who had both baseline and at least 1 follow-up patient reported outcome (PRO) assessment before treatment discontinuation.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 57 | 55
units on a scale
  Global health status / QOL | 2.82 [-1.49 to 7.13] | 2.69 [-1.70 to 7.08]
  Functional scale: Physical functioning | 0.74 [-3.26 to 4.73] | -0.46 [-4.59 to 3.66]
  Functional scale: Role functioning | -0.41 [-5.91 to 5.09] | -1.60 [-7.28 to 4.08]
  Functional scale: Emotional functioning | 4.16 [0.13 to 8.18] | 3.56 [-0.57 to 7.69]
  Functional scale: Cognitive functioning | -1.47 [-5.14 to 2.21] | -1.23 [-5.06 to 2.59]
  Functional scale: Social functioning | 1.24 [-4.43 to 6.90] | 2.08 [-3.76 to 7.92]
  Symptom scale/item: Fatigue | -2.79 [-7.04 to 1.46] | -5.12 [-9.50 to -0.75]
  Symptom scale/item: Nausea and vomiting | -0.87 [-2.63 to 0.90] | -1.04 [-2.82 to 0.74]
  Symptom scale/item: Pain | -5.98 [-11.06 to -0.90] | -6.10 [-11.32 to -0.87]
  Symptom scale/item: Dyspnoea | 3.07 [-2.15 to 8.30] | 5.09 [-0.27 to 10.45]
  Symptom scale/item: Insomnia | -4.62 [-10.33 to 1.08] | -5.02 [-10.88 to 0.84]
  Symptom scale/item: Appetite loss | 2.25 [-3.89 to 8.38] | -0.69 [-7.04 to 5.67]
  Symptom scale/item: Constipation | -4.12 [-10.30 to 2.06] | -1.33 [-7.72 to 5.07]
  Symptom scale/item: Diarrhoea | 4.26 [1.34 to 7.17] | 1.74 [-1.24 to 4.73]
  Symptom scale/item: Financial difficulties | -5.26 [-11.61 to 1.10] | -0.27 [-6.83 to 6.29]

9. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Head and Neck Module35 (EORTC QLQ-H&N35)
Description: The EORTC QLQ-H&N35 is designed to be used together with the core QLQ-C30. The recall period for the items in the module was "the past week". Items hn1 to hn30 were scored on 4 point Likert type categorical scales ("not at all", "a little", "quite a bit", "very much"). Items hn31 to hn35 had a "no/yes" response format. The scores were transformed into 0 to 100 scales, with a high score implying a high level of symptoms.Negative changes from baseline indicate deterioration in functioning / global QoL scales and improvement in symptom scales.
Time Frame: Baseline up to PCD (about 34 months)
Population: The analysis population included all ITT participants, who had both baseline and at least 1 follow-up PRO assessment before treatment discontinuation.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 57 | 55
units on a scale
  Symptom scale/item: Pain | -3.57 [-8.56 to 1.43] | -0.41 [-5.54 to 4.73]
  Symptom scale/item: Swallowing | -4.34 [-8.79 to 0.10] | -1.47 [-6.03 to 3.09]
  Symptom scale/item: Senses problems | -1.58 [-7.22 to 4.05] | -1.88 [-7.72 to 3.96]
  Symptom scale/item: Speech problems | -4.54 [-9.21 to 0.13] | -2.69 [-7.51 to 2.13]
  Symptom scale/item: Trouble with social eating | -5.55 [-10.14 to -0.96] | -0.71 [-5.42 to 4.01]
  Symptom scale/item: Trouble with social contact | -1.27 [-5.68 to 3.15] | 3.45 [-1.14 to 8.04]
  Symptom scale/item: Less sexuality | -3.32 [-11.44 to 4.80] | 4.90 [-3.72 to 13.53]
  Symptom scale/item: Teeth | -1.59 [-8.91 to 5.74] | -1.88 [-9.29 to 5.53]
  Symptom scale/item: Opening mouth | 0.35 [-5.29 to 5.99] | 0.22 [-5.56 to 5.99]
  Symptom scale/item: Dry mouth | -6.30 [-10.50 to -2.10] | 3.44 [-0.82 to 7.71]
  Symptom scale/item: Sticky saliva | -3.91 [-9.70 to 1.88] | 4.68 [-1.22 to 10.58]
  Symptom scale/item: Coughing | -3.99 [-8.67 to 0.69] | -1.72 [-6.48 to 3.04]
  Symptom scale/item: Felt ill | 1.320 [-4.22 to 6.86] | 0.12 [-5.45 to 5.70]
  Symptom scale/item: Pain killers | -13.18 [-24.49 to -1.88] | -11.39 [-23.02 to 0.24]
  Symptom scale/item: Nutritional supplements | 0.351 [-7.19 to 7.89] | -4.37 [-12.23 to 3.49]
  Symptom scale/item: Feeding tube | -6.36 [-9.58 to -3.15] | -0.11 [-3.30 to 3.08]
  Symptom scale/item: Weight loss | -17.72 [-27.23 to -8.21] | -9.47 [-19.16 to 0.22]
  Symptom scale/item: Weight gain | -3.03 [-10.08 to 4.02] | 5.16 [-1.96 to 12.27]

10. Secondary Outcome: Summary of PFS and OS for P16 Negative (%Positive Tumor Cells < 70%)
Description: A central test was defined as the tumor tissue-based p16 IHC test performed at a central laboratory (Ventana). The analysis of concordance between HPV status as assessed by local or central laboratory included the number and percentage of participants with p16 detected or not detected at the central laboratory, given that all local testing must have been negative for HPV in order for the patient to be eligible for the study. Initial analysis of the p16 status was based on the conventional cutoff of 70% p16-positive tumor cells to call out cases that might be considered HPV-positive. P16 expression was scored as positive if strong and diffuse nuclear and cytoplasmic staining was present in at least 70% of the tumor cells.
Time Frame: Screening
Population: The analysis population included all participants treated with cetuximab in combination with placebo or palbociclib who had at least 1 baseline biomarker assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 54 | 48
months
  PFS | 3.7 [3.2 to 5.6] | 5.0 [3.3 to 7.2]
  OS | 9.9 [7.1 to 13.9] | 8.0 [7.0 to 14.7]

11. Secondary Outcome: Summary of PFS and OS Based on Investigator Assessment by Rb Expression >= 1%
Description: Rb expression in the palbociclib and cetuximab treatment group, the relationship of the biomarker (individually) with PFS and OS were explored using graphical methods such as box plots, at baseline. The tumors of participants were Rb-positive, which was defined by Rb IHC with>=1% positive tumor cells.
Time Frame: Screening
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 57 | 53
months
  PFS | 3.9 [3.5 to 6.2] | 4.6 [2.6 to 5.6]
  OS | 10.5 [7.1 to 15.6] | 7.8 [6.9 to 11.8]

12. Secondary Outcome: Trough Plasma Concentration (Ctrough) and Within-participant Mean Steady-state Pre-dose Concentration (WPM-Ctrough) at Steady State for Palbociblib
Description: Ctrough is steady-state pre-dose concentration, which was observed directly from data. WPM-Ctrough is within-participant mean steady-state pre-dose concentration. For palbociclib, a steady-state trough was to be defined as a pre-dose plasma concentration following at least 7 consecutive days of 125 mg daily dose without dosing interruption and the time window for the PK collection was to be between 24 hr +/- 2 hr and 24 min post-dose the day prior to PK collection and no more than 1 hr post-dose on the day of PK collection.
Time Frame: Pre-dose of Day 15 in Cycle 1 and Cycle 2
Population: The analysis population included all as-treated participants, who were treated with the study treatments and had at least measured plasma concentration for at least 1 analyte (palbociclib and/or cetuximab)
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/ml)
Arm/Group | Palbociclib + Cetuximab
Number analyzed (Participants) | 57
nanograms per milliliter (ng/ml)
  Ctrough Cycle 1 Day 15: number analyzed (Participants) | 27
  Ctrough Cycle 1 Day 15 | 69.8 (28.208)
  Ctrough Cycle 2 Day 15: number analyzed (Participants) | 28
  Ctrough Cycle 2 Day 15 | 67.8 (28.905)
  WPM-Ctrough: number analyzed (Participants) | 37
  WPM-Ctrough | 71.6 (30.183)

13. Secondary Outcome: Ctrough and Cendinf, WPM-Ctrough and WPM-Cendinf at Steady State for Serum Cetuximab
Description: Ctrough is steady-state pre-dose concentration. Cendinf is steady-state end-of-infusion concentration. Ctrough and Cendinf were observed directly from data. WPM-Ctrough and WPM-Cendinf are within-participant mean steady-state pre-dose concentration and end-of-infusion concentration. Acceptance criteria for a steady-state Cendinf was defined as a PK sample that was 1) collected after at least 3 consecutive weeks of cetuximab IV infusions without interruption or prior dose reduction and 2) was collected at the end of cetuximab infusion time +/- 10% of the actual duration of the cetuximab infusion.
Time Frame: Pre-dose and end-of infusion of Day 15 in Cycle 1 and Cycle 2
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
Number analyzed (Participants) | 57 | 57
ng/ml
  Ctrough Cycle 1 Day 15: number analyzed (Participants) | 51 | 52
  Ctrough Cycle 1 Day 15 | 39706.4 (92) | 42914.1 (62)
  Ctrough Cycle 2 Day 15: number analyzed (Participants) | 43 | 43
  Ctrough Cycle 2 Day 15 | 51005.3 (74) | 52995.7 (71)
  WPM-Ctrough: number analyzed (Participants) | 54 | 56
  WPM-Ctrough | 45605.9 (83) | 46796.5 (63)
  Cendinf Cycle 1 Day 15: number analyzed (Participants) | 43 | 40
  Cendinf Cycle 1 Day 15 | 145748.3 (43) | 137185.5 (61)
  Cendinf Cycle 2 Day 15: number analyzed (Participants) | 37 | 41
  Cendinf Cycle 2 Day 15 | 149155.7 (38) | 153310.1 (39)
  WPM-Cendinf: number analyzed (Participants) | 46 | 50
  WPM-Cendinf | 149119.2 (36) | 148063.3 (39)

ADVERSE EVENTS:
Time Frame: From the first dose through and including 28 calendar days after the last administration of the study treatment (up to 6.9 years)
Description: The same event may appear as both an AE and a SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Arm/Group | Palbociclib + Cetuximab | Placebo + Cetuximab
All-Cause Mortality (participants affected / at risk) | 52/64 | 43/60
Serious Adverse Events (participants affected / at risk) | 25/64 | 19/60
Other Adverse Events (participants affected / at risk) | 55/64 | 53/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Cetuximab (N=64) | Placebo + Cetuximab (N=60)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Disease progression (General disorders) | 7 | 6
General physical health deterioration (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Coma (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Palbociclib + Cetuximab (N=64) | Placebo + Cetuximab (N=60)
Anaemia (Blood and lymphatic system disorders) | 23 | 8
Leukopenia (Blood and lymphatic system disorders) | 13 | 0
Lymphopenia (Blood and lymphatic system disorders) | 7 | 1
Neutropenia (Blood and lymphatic system disorders) | 19 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Constipation (Gastrointestinal disorders) | 7 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 5
Dysphagia (Gastrointestinal disorders) | 9 | 5
Nausea (Gastrointestinal disorders) | 8 | 6
Stomatitis (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 5 | 7
Fatigue (General disorders) | 8 | 8
Pyrexia (General disorders) | 9 | 8
Paronychia (Infections and infestations) | 2 | 8
Pneumonia (Infections and infestations) | 4 | 6
Alanine aminotransferase increased (Investigations) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 4
Blood creatinine increased (Investigations) | 5 | 3
Neutrophil count decreased (Investigations) | 9 | 0
Platelet count decreased (Investigations) | 10 | 0
Weight decreased (Investigations) | 5 | 3
White blood cell count decreased (Investigations) | 11 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 6 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 11 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 4
Dizziness (Nervous system disorders) | 3 | 6
Headache (Nervous system disorders) | 6 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 14 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 27 | 21
Hypertension (Vascular disorders) | 5 | 2
Hypotension (Vascular disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/20/NCT02499120/Prot_001.pdf
  • Statistical Analysis Plan (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT02499120/SAP_000.pdf